CLINICAL TRIAL: NCT03373682
Title: Safety and Efficacy of Extracorporeal Shock Wave Lithotripsy for Geriatric Patients With Chronic Pancreatitis
Brief Title: Safety and Efficacy of ESWL for Geriatric Patients With Chronic Pancreatitis
Acronym: ESWL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept., Changhai Hospital
Other Study IDs: ESWL-01
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Chronic Pancreatitis; Geriatric; Extracorporeal Shock Wave Lithotripsy
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Pancreatic extracorporeal shock wave lithotripsy (P-ESWL) is recommended as the first-line treatment for pancreatic stones. However, how well P-ESWL performs in geriatric patients remains unclear. The investigators aimed to evaluate the safety and efficacy of P-ESWL for geriatric patients with chronic pancreatitis.

DETAILED DESCRIPTION:
This prospective observational study was conducted in patients with painful chronic pancreatitis who underwent P-ESWL. Patients aged over 65 years were included in the geriatric group; patients aged under 65 years who underwent P-ESWL in the same period were assigned to the control group. For investigation of long-term follow-up, the geriatric group were matched with patients from the control group in a 1:1 ratio. The primary outcomes were P-ESWL complications and pain relief. The secondary outcomes included: stone clearance, physical and mental health, quality of life score, and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful chronic pancreatitis and radiopaque stones of ≥5mm.

Exclusion Criteria:

* Patients with a suspected or established malignant mass or pancreatic ascites, and pregnant patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic pancreatitis patients with pancreatic stones in China
Sampling Method: Probability Sample
Enrollment: 1404 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
P-ESWL complications | April 30, 2016
  The complications after P-ESWL. Including post-ESWL pancreatitis, bleeding, infection, steinstrasse, and perforation. The degree of these complications will also be measured.
Pain relief by the end of follow-up period | April 30, 2018
  Participants will be followed up annually either by return visit or telephone call. Condition of abdominal pain or acute pancreatitis attack during follow-up will be measured. Pain relief at the end of the follow-up period was classified as complete relief (Izbicki pain score≤10) or partial relief (Izbicki pain score >10 after a decrease of >50%)

SECONDARY OUTCOMES:
Stone clearance as assessed by ERCP performed post-ESWL | April 30, 2016
  Stone clearance was evaluated at the ERCP performed post-ESWL, with complete clearance defined as clearance of >90% of the main pancreatic duct stone volume, whereas partial clearance was defined as clearance of 50%-90% of the stone volume.
Physical and mental health assessed by SF-36 questionnaire | April 30, 2018
  Physical and mental health after treatment were assessed according to the scores on the SF-36 questionnaire.
Quality of life score assessed by the patient | April 30, 2018
  Quality of life score after treatment were assessed by the patient and ranged from 0 to 100, with higher scores indicating a better quality of life.
Body weight | April 30, 2018
  Body weight after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

REFERENCES:
- [Background] Wang D, Bi YW, Ji JT, Xin L, Pan J, Liao Z, Du TT, Lin JH, Zhang D, Zeng XP, Ye B, Zou WB, Chen H, Xie T, Li BR, Zheng ZH, Li ZS, Hu LH. Extracorporeal shock wave lithotripsy is safe and effective for pediatric patients with chronic pancreatitis. Endoscopy. 2017 May;49(5):447-455. doi: 10.1055/s-0043-104527. Epub 2017 Apr 12. PMID 28403504
- [Background] Hu LH, Ye B, Yang YG, Ji JT, Zou WB, Du TT, Hao JF, Jiang YY, Liao Z, Li ZS. Extracorporeal Shock Wave Lithotripsy for Chinese Patients With Pancreatic Stones: A Prospective Study of 214 Cases. Pancreas. 2016 Feb;45(2):298-305. doi: 10.1097/MPA.0000000000000464. PMID 26418906
- [Background] Li BR, Liao Z, Du TT, Ye B, Chen H, Ji JT, Zheng ZH, Hao JF, Ning SB, Wang D, Lin JH, Hu LH, Li ZS. Extracorporeal shock wave lithotripsy is a safe and effective treatment for pancreatic stones coexisting with pancreatic pseudocysts. Gastrointest Endosc. 2016 Jul;84(1):69-78. doi: 10.1016/j.gie.2015.10.026. Epub 2015 Nov 2. PMID 26542375
- [Background] Li BR, Liao Z, Du TT, Ye B, Zou WB, Chen H, Ji JT, Zheng ZH, Hao JF, Jiang YY, Hu LH, Li ZS. Risk factors for complications of pancreatic extracorporeal shock wave lithotripsy. Endoscopy. 2014 Dec;46(12):1092-100. doi: 10.1055/s-0034-1377753. Epub 2014 Sep 24. PMID 25251205